CLINICAL TRIAL: NCT05281224
Title: Ventilator Tube Holder for Patients With a Tracheostomy: A Pilot Usability Study Protocol
Brief Title: Ventilator Tube Holder for Patients With a Tracheostomy
Acronym: TRACHVest
Status: Completed | Type: Observational
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Other Study IDs: CED211
Record Dates: First submitted 2021-11-30; First posted 2022-03-16 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-03

CONDITIONS: Critical Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients admitted to the critical care unit (CCU) at University Hospital Wales (UHW) have a variety of life-threatening conditions which require specialist care, often including a period of sedation and mechanical ventilation. As a consequence of critical illness, survivors often experience multiple sequela, including muscle weakness which leads to reduced mobility and physical function, especially if they experience a prolonged stay within critical care. Patients who require mechanical ventilation (MV) usually initially receive this via an endotracheal tube (ETT), but if the need for MV continues then this support is delivered through a tracheostomy tube. A small opening is made in the front of the patient's neck and the tracheostomy tube inserted into the trachea. This is connected to the ventilator and allows ventilatory support to be delivered without the need for an ETT. Consequently, sedation levels can be reduced, facilitating improved patient comfort, communication, eating, drinking and mobilisation.

Early rehabilitation is a key component of a patient's critical care journey and patients are supported with this by a number of specialist staff including physiotherapists, occupational therapists, nurses and support workers. Part of this rehabilitation may include helping a patient to sit on the edge of the bed, stand and mobilise. During rehabilitation sessions and other aspects of patient care, safety is paramount and staff must take care to ensure all lines and attachments are not dislodged. This includes tubing connecting the ventilator to the tracheostomy, excessive movement of which can cause damage to the airway, breakdown of skin and partial or complete dislodgement requiring immediate intervention.

The number of staff required to help mobilise a patient and maintain safety can be significant, especially when the patient has several attachments. Unfortunately, this staffing burden may contribute to reduced levels of patient mobilization and rehabilitation. However, it is possible that specially designed equipment may facilitate patient mobilization with increased safety and reduced resource requirements. This study will test a garment that may achieve this and obtain staff and patient opinion on its utility.

DETAILED DESCRIPTION:
Patient A was an 85-year-old female with motor neurone disease and a permanent tracheostomy. She was dependent on a respiratory ventilator, but relatively mobile within the critical care unit. However, the ventilator tubing connecting the ambulatory ventilator (usually located behind the patient) to the tracheostomy interfered with the patient's freedom to move and disturbed the tracheostomy as she changed position. A custom-made garment was designed by the Medical Engineering Department of Cardiff and Vale University Health Board (CVUHB) to hold the tubing still and out of the way. This relieved any pressure or pulling on the tracheostomy tube and allowed the patient greater freedom of movement without requiring additional staff to manage/handle the tubing. Patient A used the garment every day for prolonged periods (2-3 hours) and for a duration of 3 months, before she became bedbound and no longer needed it.

The apparent success of this custom-made garment could be repeated in other patients with similar conditions. Furthermore, it may help to reduce the number of staff required when mobilising a patient and lower the handling burden. This project is intended to explore the use of such a garment in a critical care setting. Patients who can be moved out of bed may be moved several times a day, requiring 3 or more staff members each time. If the garment holds the connector tubing securely during these movements then there are several potential benefits:

* Fewer staff may be required to move the patient
* Improved manual handling processes for staff
* Reduction in adverse events associated with mobilisation
* Improved patient comfort during mobilisation Even small movements of the tracheostomy tube can cause discomfort and coughing, whereas larger movements risk tissue damage, airway trauma or dislodging the tracheostomy. In addition, the patient may have more freedom of movement when using the garment out of bed.

However, it is uncertain if or how the current design of the garment will impact on staff and patient activities. There are several potential disadvantages of using the garment:

* It may be awkward to put on and take off, especially for patients with multiple device connections and/or cannulas, limited upper body mobility, and/or cognitive impairment
* It may interfere with the use of a hoist
* As a result, it may increase the time and/or staff members needed to move the patient
* It may increase motion of the tracheostomy tube resulting in greater discomfort and risk of tissue damage or disruption of the ventilation
* It may be uncomfortable or too hot for the patient
* Staff may become dependent on the garment and be less vigilant of the tubing. Essentially, the study will observe staff using the garment to determine where the potential benefits and limitations exist.

ELIGIBILITY:
Inclusion Criteria:

- Inpatient on critical care unit for any admitting condition

* Aged over 18
* Any gender
* A permanent or temporary tracheostomy
* Dependant on a respiratory ventilator
* Capable and expected to be out of bed and mobile on the critical care unit with the assistance of staff
* Expected to remain on critical care unit for several days, and to retain their tracheostomy during this time.
* Not currently Covid-positive (defined by local policy) and in area of reduced requirement for personal and protective equipment
* Is able to give written, informed consent or have an appropriate consultee who can be approached

Exclusion Criteria:

* Injuries or restricted movement of the arms or shoulders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical care
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Staff opinion on potential to change occurrence of adverse events using TrachVest | 6 months
  User feedback via questionnaires and focus groups to determine its potential to reduce adverse events. Questionnaires will be non-validated. Focus groups to follow structured questions.

SECONDARY OUTCOMES:
Perceived benefits of the TrachVest on staff time | 6 months
  User feedback via questionnaires and focus groups to determine its potential to reduce staff time. Questionnaires will be non-validated for staff and patients. Staff focus groups to follow structured questions.
Perceived benefits of the TrachVest on patient comfort | 6 months
  User feedback via questionnaires and focus groups to determine its potential to improve patient comfort. Questionnaires will be non-validated for staff and patients. Staff focus groups to follow structured questions.
Usability of the TrachVest | 6 months
  User feedback via questionnaires and focus groups to determine its usability within critical care. Questionnaires will be non-validated for staff and patients. Staff focus groups to follow structured questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and Vale UHB, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No